CLINICAL TRIAL: NCT01093209
Title: Efficacy of the Interferential Laser Therapy in Pain Reduction in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: EFFICACY OF THE INTERFERENTIAL LASER THERAPY IN THE REDUCTION OF PAIN IN CARPAL TUNNEL SYNDROME., Hospital Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ramón y Cajal Hospital
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-03

CONDITIONS: Carpal Tunnel Syndrome; Neuropathic Pain
Keywords: Carpal Tunnel Syndrome; Interferential laser therapy; Low-level laser therapy; Neuropathic pain; Median nerve compression
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Laser Therapy (Sham Comparator)
  Interventions: Device: Interferential Laser Therapy
- Interferential Laser Therapy (Active Comparator)
  Interventions: Device: Interferential Laser Therapy

INTERVENTIONS:
Device: Interferential Laser Therapy — PROCEDURE: Interventional group: Two independents and identical probes. Energy dose per point and per probe: 5 J. Continuous emission. Treatment time:8 minutes. Sessions: 10. Frequency of the sessions: daily. Irradiation technique: handily, in contact and at 7 points over distal pathway of median nerve.Control group: Sham laser:650 nm.Scanning mode.Outpout power:1 mW.

SUMMARY:
The purpose of this study is to determine the efficacy of the interferential laser therapy in the wrist and hand pain and disability reduction and force improvement in the carpal tunnel syndrome. Subjects are patients diagnosed of carpal tunnel syndrome who have been prescribed laser therapy. Settings: Ramon y Cajal Hospital. Department of Rehabilitation. Physical therapy unit. Electrotherapy section. Occupational Therapy. Department of Neurology.

DETAILED DESCRIPTION:
The spatiotemporal superposition of two independent and opposite beams of laser generates a constructive interference pattern that increases the therapeutic effects in the irradiated tissue. Patient suffering pain from diagnosed carpal tunnel syndrome will receive conventional or interferential laser therapy. This is a comparative randomized and double blind clinical study. Two identical lasers in near infrared range will be used. Frequency of sessions: daily. Irradiated technique: manual, contact and punctual. Pain will be evaluated by visual analog scale at rest and during analytical wrist movement. Disability will be evaluated by the DASH and BOSTON questionnaire. Evaluation will take place at pre and post-treatment times.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of Carpal Tunnel Syndrome by means of an Electromyography Study.
* Patients with or not previous surgery.
* Patients with an age of 18 years or older.
* Patients having a signed informed consent.

Exclusion Criteria:

* Patients with severe hand traumatisms.
* Patients with cervical radiculopathy.
* Patients with Outlet Thoracic Syndrome.
* Patients bearing osteo syntheses material.
* Patients suffering tumoral pathology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 5 minutes
  Visual Analogue Scale during wrist analitical movements.

SECONDARY OUTCOMES:
Disability Arm Shoulder and Hand questionnaire (DASH) | 15 minutes
Boston Carpal Tunnel Questionnaire | 5 minutes
Dinamometry | 5 minutes
  Power grip and pinch grip.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Montes-Molina, PT, MsC, Principal Investigator — Unit of Physiotherapy; Fidel Martinez-Ruiz, Physicist, Study Director — Unit Biomechanics and Biomaterials
Locations (1):
- Ramón y Cajal University Hospital, Madrid, Madrid, Spain